CLINICAL TRIAL: NCT06330857
Title: Evaluation of Anatomy and Symptoms After Surgery With a Novel Anterior Rectopexy in a Cohort With Combined Pelvic Defects.
Brief Title: Recurrence and Bowel Function After Laparoscopic Vaginorectopexy, a Modified Anterior Rectopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bjarne Melvas, Consultant, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr2021-06921-02
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Rectal Prolapse; Fecal Incontinence; Defecation Disorder; Enterocele; Rectocele
Keywords: laparoscopy; obstructive defecation
MeSH Terms: conditions — Rectal Prolapse; Fecal Incontinence; Hernia; Rectocele

STUDY DESIGN:
Intervention Model Description: Evaluation of recurrence with clinical examination and defecography. Evaluation of bowel function with a questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical intervention (Experimental): Operated with the intervention, ie vaginorectopexy
  Interventions: Procedure: Laparoscopic vaginorectopexy

INTERVENTIONS:
Procedure: Laparoscopic vaginorectopexy — Modified laparoscopic anterior rectopexy for multiple pelvic prolapses

SUMMARY:
Several pelvic prolapses can render defecation difficulties and they are often treated with different surgical techniques. This study will evaluate a novel variation of a laparoscopic technique used to treat rectal prolapse that is modified to treat multiple pelvic prolapses. 25 women with symptoms of obstructed defecation and multiple pelvic prolapses are assessed before and after surgery with clinical examination, defecography and a questionnaire for bowel function and quality of life. Follow up was scheduled after three and twelve months and at long term (minimum ten years).

DETAILED DESCRIPTION:
Patients and Methods

Patients From 2002 to 2008, referred patients with symptoms of obstructed defecation (=OD) and diagnosed with multiple posterior pelvic organ prolapse (=PPOP) (protocol below) were considered for inclusion in the study. More than one defect (internal-or external rectal prolapse, Enterocele (EC) or Rectocele (RC)) was denoted as multiple PPOP. Patients were evaluated with clinical examination, defecography and a questionnaire that evaluated bowel function and bowel-related quality of life (QoL). Patients who did not respond to conservative treatment (diet advice, oral bulking agents, rectal enemas and/or bio-feedback) were offered inclusion in the study.

Patients with anismus were excluded after evaluation with a combination of defecography (see below) and manometry.

Surgical procedure Pneumoperitoneum was established with Verres needle. Two 12 mm trocars are placed at the umbilicus and two cm above the symphysis. Two 5 mm trocars are placed in the right and left iliac fossa. The procedure starts with an incision exposing the promontory which continues down along the right peritoneal reflection (Fig 9). A limited dissection of the promontory and a shallow unilateral incision was employed to avoid damage to the superior hypogastric plexus and the hypogastric nerves. The rectovaginal space was opened down to the pelvic floor, exposing the pelvic floor muscles. A T-shaped Vypro-mesh was inserted into the rectovaginal space and sutured to the pelvic floor muscles lateral to the vagina and to the distal vagina with a non-absorbable suture (EthibondR,). Two additional sutures fixated the mesh to the sacrouterine ligaments, closing the rectovaginal space and elevating the pouch of Douglas. Staples were used to anchor the mesh to the promontory as well as the mesorectum to the mesh, preventing rectal intussusception. The peritoneal defect was closed with a running, absorbable suture.

Bowel Function Questionnaire The symptom load was evaluated with Linkoping Bowel function Questionnaire (LBQ). It is a quantitative bowel function questionnaire that evaluates four domains: fecal incontinence, constipation, OD and bowel-related quality of life. Symptom load is graded in four levels. Questions considered most relevant for each category of OD, incontinence and QoL were used for the longitudinal analyses.

Defecography

The defecography used plain X-ray and pictures/film were recorded at rest and during straining with the patient situated on a commode. Preparations included oral, rectal and vaginal contrast. Examination of the investigation was made by two senior radiologists and the following protocol was used for evaluation:

Rectal prolapse Oxford grading system 1-5 for intususception and external prolapse.

Enterocele Grade1 EC reaching below cervix, but not distal to half of the vaginal length. Grade 2 EC reaching below half of the vaginal length, but not below the sphincter plane.

Grade 3 EC protruding below the sphincter plane and out of the anal canal.

Rectocele A protrusion beyond the imaginary line between the sphincter and the rectum over or equal to 2 cm in depth.

Anismus The inability to open the anal canal during evacuation of rectal contrast without an anatomical reason. The puborectal function is evaluated separately regardless of signs of anismus with assessment of the anorectal angle.

The following protocol was used at follow-up visits:

3 months: Recording of per -and postoperative complications. Review of medical records and visit at the outpatient clinic.

12 months:

1. Clinical examination by one surgeon and one gynaecologist
2. Defecography
3. Bowel function questionnaire (LBQ)

Since defecographic evaluation was not always available due to technical failure and/or patient related factors, the evaluation protocol was adjusted according to the reliability of the clinical examination. Clinical evaluation of EC and internal prolapse (IRP) is difficult and unreliable. However, clinical evaluation of RC (> 2cm), is considered reliable. Therefore, clinical evaluation was considered sufficient for evaluation of rectocele, but not for enterocele or internal prolapse.

The following protocol was used:

Rectal prolapse and RC: Clinical evaluation and defecography. If defecography was not evaluable, clinical evaluation was considered sufficient.

IRP and EC: Clinical evaluation and defecography. If defecography was not evaluable, clinical evaluation was considered insufficient.

Long term:

During 2020, LBQ was sent to all patients who were alive achieving a minimum of 10 years follow-up; patients who did not respond were contacted via telephone. Median follow-up was 16 years (10-18 years)

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of obstructed defecation, more than one posterior pelvic organ prolapse, undergone conservative treatment

Exclusion Criteria:

* Anismus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-05-28 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Recurrence | One year
  Clinical and radiological assesment of relapse of prolapse
Bowel function | Over ten years
  Questionnaire regarding fecal incontinence and obstructed defecation
Bowel related quality of life | Over ten years
  Questionnaire regarding bowel related quality of life

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Complications within 30 days after surgery
Peroperative complications | surgery
  Complications during surgery
Operative time | minutes
  Time from start of operative procedure to the end of surgery
Conversions to open surgery | Numbers
  Numbers of operations where conversion to open surgery were necessary
Hospital days | days
  Number of days in hospital after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lars Borjesson, Professor, Principal Investigator — Göteborg University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mellgren A, Bremmer S, Johansson C, Dolk A, Uden R, Ahlback SO, Holmstrom B. Defecography. Results of investigations in 2,816 patients. Dis Colon Rectum. 1994 Nov;37(11):1133-41. doi: 10.1007/BF02049817. PMID 7956583
- [Background] D'Hoore A, Penninckx F. Laparoscopic ventral recto(colpo)pexy for rectal prolapse: surgical technique and outcome for 109 patients. Surg Endosc. 2006 Dec;20(12):1919-23. doi: 10.1007/s00464-005-0485-y. PMID 17031741
- [Background] van Geluwe B, Wolthuis A, Penninckx F, D'Hoore A. Lessons learned after more than 400 laparoscopic ventral rectopexies. Acta Chir Belg. 2013 Mar-Apr;113(2):103-6. PMID 23741928
- [Background] Mellgren A, Dolk A, Johansson C, Bremmer S, Anzen B, Holmstrom B. Enterocele is correctable using the Ripstein rectopexy. Dis Colon Rectum. 1994 Aug;37(8):800-4. doi: 10.1007/BF02050145. PMID 8055725
- [Background] Boons P, Collinson R, Cunningham C, Lindsey I. Laparoscopic ventral rectopexy for external rectal prolapse improves constipation and avoids de novo constipation. Colorectal Dis. 2010 Jun;12(6):526-32. doi: 10.1111/j.1463-1318.2009.01859.x. Epub 2009 Apr 10. PMID 19486104
- [Background] Tsunoda A, Takahashi T, Matsuda S, Kusanagi H. Long-term annual functional outcome after laparoscopic ventral rectopexy for rectoanal intussusception and/or rectocele: evaluation of sustained improvement. Tech Coloproctol. 2021 Dec;25(12):1281-1289. doi: 10.1007/s10151-021-02499-4. Epub 2021 Oct 11. PMID 34633567